CLINICAL TRIAL: NCT02476903
Title: Viscosupplementation in the Hip Following Hip Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: Sean McMillan, DO (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2015Salvo
Record Dates: First submitted 2015-06-17; First posted 2015-06-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid

INTERVENTIONS:
Drug: Monovisc

SUMMARY:
Hip arthroscopy is a rapidly evolving procedure that has seen an exponential increase in the number of cases performed yearly. With hip arthroscopy still in its infancy in relation to knee and shoulder arthroscopy, there are still many questions yet to be answered. Axioms that were once thought to be true regarding indications and treatment for hip arthroscopy are continually being revised. As with the knee and shoulder before it, the hip is now graduating into treatment avenues that were otherwise thought to only be possible through an open surgical procedure.

Viscosupplementation in patients post arthroscopy with known articular cartilage injury has been shown to be efficacious. The pathophysiology of hyaline degradation during the arthritic process within the knee has been studied, and with this understanding has grown the widespread usage of viscosupplementation. While questions still exist regarding the effectiveness of viscosupplementation in non-weightbearing joints, it appears the benefits seen in the weight bearing joints, such as the knee, are apparent

ELIGIBILITY:
Inclusion Criteria:

Preoperative inclusion criteria will be made via x-ray and MRI evaluation. These criteria shall include: 2 mm or greater joint space preservation of the hip on radiographs, absence of acetabular subcortical bone cysts, Tonnis Score less than 2 on radiographs, and patient age greater than 18.4 Intra-operative evaluation of the cartilage will be performed by the surgeon on both the acetabular and femoral head sides. Patients shall be included if the osteochondral defect meets Outerbridge Classification criteria of stage II or greater. Furthermore the lesion shall be greater than 1cm in size (and thus not amenable to other procedures such as microfracture). Subjects must be willing to sign the IRB-approved informed consent and be older than 18 years old.

Exclusion Criteria:

All patients 55 years of age and older. All patients with previous hip surgery on a concomitant side. Patients who present a history of radiculopathy or regional pain syndrome. Patients with a worker's compensation claim or pending litigation claim. Patients with Outerbridge Grade IV changes on either acetabular or femoral articular cartilage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Pain Using Visual Analog Scale | Up to 12 months
  Using Visual Analog Scale